CLINICAL TRIAL: NCT00002285
Title: A Phase I/II Pilot Trial To Evaluate Zidovudine (AZT) and T Lymphocyte Transfer in the Treatment of Human Immunodeficiency Virus Type-III (HIV) Infection in AIDS Patients
Brief Title: A Study of Zidovudine and T Lymphocyte Transfer in the Treatment of HIV Type III in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 014B; 27433-10
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: HIV Infections
Keywords: Virus Replication; Pilot Projects; Immune Tolerance; Lymphocytes; Drug Evaluation; Combined Modality Therapy; Acquired Immunodeficiency Syndrome; Transplantation, Homologous; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine the safety and efficacy of zidovudine (AZT) treatment combined with syngeneic or HLA identical allogeneic lymphocyte transfer in the presence of interleukin 2 (IL-2) as a treatment for AIDS. Patients with documented HIV viremia will be evaluated. Effects on virus replication, immune function, and clinical condition will be monitored with periodic virus cultures, estimates of lymphocyte type and numbers, cell surface markers, in vitro lymphocyte responses and frequent clinical evaluations.

ELIGIBILITY:
Inclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

- Lymphoma. Active central nervous system (CNS) infection by bacteria, varicella zoster virus, herpes simplex virus, or Cryptococcus neoformans. Any prior CNS infection due to Toxoplasma gondii. Any active life-threatening infection including Pneumocystis carinii pneumonia (PCP) (if prior PCP then pre-PCP arterial PO2 must be above 80), disseminated cryptococcosis (if there was a prior cryptococcosis infection the patient must have had a negative blood and cerebrospinal fluid (CSF) culture taken more than 6 weeks after the last antifungal therapy).

Any prior mycobacterium avium-intracellulare isolation.

Patients with the following conditions are excluded:

- Lymphoma. Active central nervous system (CNS) infection by bacteria, varicella zoster virus, herpes simplex virus, or Cryptococcus neoformans. Any prior CNS infection due to Toxoplasma gondii. Any active life-threatening infection including Pneumocystis carinii pneumonia (PCP) (if prior PCP then pre-PCP arterial PO2 must be above 80), disseminated cryptococcosis (if there was a prior cryptococcosis infection the patient must have had a negative blood and cerebrospinal fluid (CSF) culture taken more than 6 weeks after the last antifungal therapy).

Any prior mycobacterium avium-intracellulare isolation. Patients accepted for allogenic cell transfer must meet the CDC criteria for AIDS. Those patients who meet the criteria only because of Kaposi's sarcoma must also have a history of generalized lymphadenopathy (CDC category III), neurologic disease (CDC category IV-B), or constitutional disease (CDC category IV-A). Patients may be accepted for syngeneic cell transfer even if they have not met the CDC AIDS criteria, provided they have had constitutional disease (CDC category IV-A) or a specified non-AIDS defining secondary infection (CDC category IV-C2).

Patients must have a positive blood culture for the AIDS virus before the beginning of therapy.

Patients must be skin test negative for PPD. Patients must have a life expectancy of at least 6 months and a Karnofsky status of 60 or above.

Patients must sign an informed consent agreement. From eligible patients precedence will be given to those with identical twin donors, then to Minnesota residents. The first patient must have an identical twin donor. Among eligible Minnesota patients without identical twin donors, the order of enrollment will be determined by overall good health, the presence of Kaposi's sarcoma (which permits monitoring of response by measuring lesions) and/or the presence of cytomegalovirus (CMV) viremia (which permits monitoring of response by remission of CMV viremia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States